CLINICAL TRIAL: NCT01273727
Title: Ozurdex in Treatment of Macular Edema Post Membrane Peeling
Brief Title: Ozurdex for Macular Edema Post Membrane Peeling
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Retina Specialists, PC (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, John Khadem, Principal Investigator, Retina Specialists, PC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3433-001
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Epiretinal Membrane; Cellophane Maculopathy; Macular Edema; Retinal Edema
Keywords: epiretinal membrane; macular pucker; cellophane maculopathy; macular edema; retinal edema; ozurdex; dexamethasone; intravitreal implant
MeSH Terms: conditions — Epiretinal Membrane; Macular Edema; Papilledema | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No Ozurdex (No Intervention): Arm 1(control) - Patients who have had epi-retinal membrane peeling and have macular edema at least 3 months (90 days) after surgery. These patients will followed without Ozurdex. The patients will be treated with current standard of care, including topical and intravitreal or subtenon's medication.
- Ozurdex 3 months after surgery (Experimental): Patients who have had epi-retinal membrane peeling and have residual macular edema 3 months after surgery. These patients will receive an Ozurdex implant
  Interventions: Drug: Dexamethasone
- Ozurdex 6 months or longer after surgery (Experimental): Patients who have had epiretinal membrane peeling and have residual macular edema at least 6 months after surgery
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — intravitreal implant 0.7 mg 6 month duration
  Other Names: Ozurdex
  Arms: Ozurdex 3 months after surgery
Drug: dexamethasone — intravitreal implant 0.7 mg duration 6 months
  Other Names: ozurdex
  Arms: Ozurdex 6 months or longer after surgery

SUMMARY:
An epiretinal membrane is scar tissue on the retina that can cause blurring and distortion of vision and lead to swelling, or macular edema. Despite surgery to remove the scar tissue(membrane peeling), residual swelling of the retina may continue to interfere with vision.

In this study the investigators will inject an implantable steroid device into the back, fluid-filled portion of the eye. Steroids have been found to decrease the swelling in the retina. Ozurdex™ is an implantable steroid. Once implanted, Ozurdex™ is slowly dissolved by the vitreous gel that fills the eye, releasing the steroid. The steroid drug delivery system in this study, known as Ozurdex™ has been FDA-approved by the US Food and Drug Administration (FDA) for decreasing swelling due to another condition in the eye. This study will help to find out whether or not this device Ozurdex™ is also effective for reducing the swelling of the retina in patients who have already had surgery to remove scar tissue on the retina.

ELIGIBILITY:
Inclusion Criteria

* Patients with macular edema who have had previous epi-retinal membrane peeling surgery for macular edema associated with epi-retinal membranes.
* All patients must have clear ocular media/lenses determined visually by the investigator in order to permit good quality stereoscopic fundus photography, fluorescein angiography and ocular coherence tomography.

Exclusion Criteria:

* Best corrected visual acuity 20/50 or better in the study eye
* Sub-macular hemorrhage in the study eye
* Sub-retinal fibrosis in the study eye
* Macular hole in the study eye
* Active inflammatory disease of the study eye
* Choroidal neovascularization in the study eye
* History of other ophthalmic disorders with the exception of cataract or previous cataract extraction in the study eye
* Active ocular infection in the study eye
* Previous subfoveal laser treatment in the study eye
* Previous verteporfin photodynamic therapy in the study eye
* Any systemic medical condition that would preclude them from undergoing surgery with monitored sedation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
mean best corrected visual acuity as measured by Snellen visual acuity compared to enrollment | 6 months

SECONDARY OUTCOMES:
mean decrease in area and or volume of central foveal thickness as measured by OCT compared to enrollment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Khadem, MD, Principal Investigator — Retina Specialists, PC
Locations (1):
- Retina Specialists PC, New York, New York, United States